CLINICAL TRIAL: NCT03328923
Title: Acute Post-prandial Cognitive Effects Following Brown Seaweed Extract
Brief Title: Effects of Seaweed Extract on Mental Performance Following a High-carbohydrate Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: innoVactiv Inc. (Industry)
Responsible Party: Principal Investigator, Crystal Haskell-Ramsay, Associate Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 46BK1
Record Dates: First submitted 2017-10-23; First posted 2017-11-01 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Cognitive Change
Keywords: post-prandial cognition; brown seaweed

STUDY DESIGN:
Intervention Model Description: Participants will receive either 500mg brown seaweed powder (InSea2) or placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 500mg brown seaweed powder (Experimental): 2 x 250mg capsules InSea2® (brown seaweed powder)
  Interventions: Dietary Supplement: 500mg brown seaweed powder
- Placebo (Placebo Comparator): 2 x capsules microcrystalline cellulose (bulking agent) (0mg InSea2®)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: 500mg brown seaweed powder
  Other Names: InSea2®
  Arms: 500mg brown seaweed powder
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The current study will explore the impact of seaweed extract on cognitive function following a high-carbohydrate meal at a number of time-points post-consumption.

DETAILED DESCRIPTION:
The current randomised, placebo-controlled, double-blind, parallel groups study will examine the impact of a brown seaweed extract (InSea2) on cognitive function post-prandially in 60 healthy non-elderly adults who self-report post-meal drowsiness. Computerised measures of episodic memory, attention and subjective state will be completed at baseline and for 3 hours following lunch with either seaweed or placebo consumed 30 minutes prior to a carbohydrate-rich meal.

ELIGIBILITY:
Inclusion Criteria:

* Report post-meal drowsiness

Exclusion Criteria:

Below 18 or above 65 years old at the time of giving consent

* Do not report post-meal drowsiness
* Any pre-existing medical condition/illness
* History of/current head trauma
* History of intestinal tract surgery
* History of/current diagnosis of drug/alcohol abuse
* Currently taking prescription medications (excluding the contraceptive pill)
* Habitual use of dietary/herbal supplements
* Learning difficulties, ADHD (attention deficit hyperactivity disorder), dyslexia
* Frequent migraines that require medication more than once/month.
* Visual impairment that cannot be corrected with glasses or contact lenses
* Smoking
* Excessive use of caffeine (>500mg per day) from all dietary sources
* Not a native English speaker
* Food intolerances/sensitivities, including seafood/fish allergy
* Pregnancy, seeking to become pregnant, or current lactation
* BMI <18.5 or >30 kg/m2
* Any health condition that would prevent fulfilment of the study requirements
* Inability to complete all of the study assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06-23 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2016-07-28 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | Change from baseline following acute treatment, measured at 50, 90, 130, 170 and 210 minutes post-dose
  Immediate word recall, simple reaction time, digit vigilance and choice reaction time measured via the Computerised Mental Performance Assessment System (COMPASS, Northumbria University)

SECONDARY OUTCOMES:
Subjective state | Change from baseline following acute treatment, measured at 50, 90, 130, 170 and 210 minutes post-dose
  Concentration, mental stamina, physical stamina, mental tiredness, physical tiredness, hunger, thirst and fullness visual analogue scales measured via the Computerised Mental Performance Assessment System (COMPASS, Northumbria University)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Haskell-Ramsay, Dr, Principal Investigator — Northumbria University

IPD SHARING:
Plan to Share IPD: No